CLINICAL TRIAL: NCT06774248
Title: Expanding the Youth Opioid Recovery Support (YORS) Intervention for MOUD Adherence to Adolescents With OUD
Acronym: YORS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Potomac Health Foundations (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R34DA062260-01 (NIH)
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use Disorder
Keywords: adolescents; addiction; concerned significant other; family therapy; Medications for opioid use disorder; medication adherence; buprenorphine; naltrexone
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive; Medication Adherence

STUDY DESIGN:
Intervention Model Description: The Youth Opioid Recovery Support (YORS) model is an innovative wrap-around approach that attempts to address barriers to medication adherence in this vulnerable adolescent population. The YORS intervention primary components are (as detailed below):
  1. Low barrier access to MOUD, including home delivery, ride-share app transportation and mobile van delivery and low barrier access to MOUD in general
  2. Engagement of families in collaborative treatment planning and monitoring with a focus on medication adherence
  3. Assertive continuing care: actively tracking and communicating with youth and families by text and social media to promote engagement and adherence
  4. Contingency management: to provide incentives for medication adherence
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Youth Opioid Recovery Support (YORS) (Experimental): All adolescent patient participants and their treatment significant other (TSO) participants will be assigned to the YORS intervention condition for 26 weeks of treatment. YORS is an innovative wrap-around approach that attempts to enhance adherence to medication for opioid use disorder (MOUD) for adolescents with OUD. The intervention will begin upon confirming eligibility and interest in the study through screening and informed consent processes. Participants will be maintained in the YORS arm and continue to receive assertive outreach in attempts to re-engage them for the duration of the intervention period unless the withdraw from the study or are otherwise removed.
  Interventions: Behavioral: Youth Opioid Recovery Support (YORS)

INTERVENTIONS:
Behavioral: Youth Opioid Recovery Support (YORS) — The Youth Opioid Recovery Support (YORS) model is an innovative wrap-around approach that attempts to address barriers to medication adherence in this vulnerable young adult population. The YORS intervention primary components are (as detailed below):
  1. Low barrier access to MOUD, including home delivery, ride-share app transportation and mobile van delivery and low barrier access to MOUD in general
  2. Engagement of families in collaborative treatment planning and monitoring with a focus on medication adherence
  3. Assertive continuing care: actively tracking and communicating with youth and families by text and social media to promote engagement and adherence
  4. Contingency management: to provide incentives for medication adherence

SUMMARY:
Despite rising rates of fatal opioid overdoses in the United States, adolescents with OUD are far less likely than adults to receive and be retained on medication for opioid use disorder (MOUD). The multicomponent Youth Opioid Recovery Support (YORS) intervention for young adults seeks to increase adherence to extended-release MOUD and reduce opioid relapse through family involvement, assertive outreach, low-barrier access to MOUD, and contingency management. By expanding investigations of the evidence based YORS intervention to adolescents, especially those on sublingual buprenorphine, this project will significantly contribute to our knowledge base of practical strategies to address the opioid crisis in youth.

DETAILED DESCRIPTION:
Adolescents with OUD are a critical but underserved population. Despite rising rates of fatal opioid overdoses in the United States, adolescents with OUD are far less likely than adults to receive and be retained on medication for opioid use disorder (MOUD). Estimates of timely MOUD initiation among adolescents with OUD are ≤ 5% and only a quarter of residential addiction treatment facilities for adolescents even offer buprenorphine. Among the few adolescents with OUD who do receive MOUD, adherence is alarmingly low.

The multicomponent Youth Opioid Recovery Support (YORS) intervention for young adults seeks to increase adherence to extended-release MOUD and reduce opioid relapse through family involvement, assertive outreach, low-barrier access to MOUD, and contingency management. This project will expand the investigation of the YORS intervention, with demonstrated efficacy in young adults, to the critical underserved population of adolescents with OUD. Adolescents are theoretically even more likely than young adults to respond to YORS components such as family involvement, persuasion, and leverage because of their developmentally normative greater reliance on parental guidance and influence. Through this project investigators also will expand the YORS intervention to include adolescents choosing sublingual buprenorphine, which are adaptations responsive to our local clinical experience and national trends.

To achieve these aims, investigators will test the feasibility and pilot impact of YORS for N=40 adolescents and their family members in an uncontrolled, single arm clinical trial in preparation for a future larger scale randomized controlled trial. Because the preferred MOUD for adolescents in our clinical experience has been daily sublingual buprenorphine (rather than XR-MOUD), investigators will adapt YORS for sublingual buprenorphine. Finally, investigators will also conduct qualitative interviews to better understand the experience of adolescents with OUD and their families.

ELIGIBILITY:
Inclusion Criteria for adolescent patients with OUD:

1. English speaking
2. Provision of signed and dated informed assent form (may be collected verbally over audio and/or video platform in the event of a remote enrollment)
3. Willing to have a legal, English-speaking guardian provide informed consent (may be collected verbally over audio and/or video platform in the event of a remote enrollment)
4. Stated willingness to comply with all study procedures and the YORS intervention
5. Age 13-21 (inclusive)
6. Documented diagnosis of opioid use disorder (OUD)
7. Presenting for an index episode of inpatient or outpatient treatment at Maryland Treatment Centers with at least one day of opioid use in the 30 days prior to enrollment
8. Considering treatment with XR-NTX, XR-BUP, or SL-BUP* OR has begun SL-BUP maintenance treatment within the past two weeks
9. Willing to designate a parent, family member, or other person to be involved in their OUD treatment as a Treatment Significant Other
10. Access to a mobile phone

Inclusion criteria for Treatment Significant Other (TS) participants

1. English speaking
2. Provision of signed and dated informed consent form (may be collected verbally over audio and/or video platform in the event of a remote enrollment)
3. Stated willingness to comply with all study procedures and the YORS intervention
4. Parent, legal guardian, or other treatment support person designated by an adolescent patient participant to be involved in their OUD treatment as a Treatment Significant Other
5. Age 18 years or older
6. Access to a mobile phone

Exclusion Criteria for adolescent patients with OUD:

1. Psychiatric or medical instability that, in the opinion of the PI, would preclude participation in the trial (e.g., suicidality, psychosis, Sickle Cell disease with frequent crises)
2. Living situation that, in the opinion of the PI, would preclude participation in the trial (e.g., location greater than 75 miles from the treatment center, homelessness)

Exclusion Criteria for Treatment Significant Other (TSO) Participants:

1. Known to currently be sharing drugs with the adolescent participant

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative MOUD exposure | 26 weeks
  Cumulative days of exposure to MOUD during study intervention period course of treatment, which is operationalized as the proportion of time on prescribed MOUD at 26-weeks compared to the period of time in the intervention.

SECONDARY OUTCOMES:
Adverse Events and Serious Adverse Events | 26 weeks
  Adverse Events and Serious Adverse Events will be tabulated and described for severity and relatedness to the intervention.
Acceptability | 26 weeks
  Quantitative scores and qualitative feedback on Treatment Satisfaction Surveys and Interviews will be summarized and described.
Participants Enrolled | 26 weeks
  Number of participants enrolled in the intervention will be tabulated
Opioid Relapse | 26 weeks
  Opioid relapse (Y/N) will amalgamate self report and urine drug screen data. Relapse is defined as 10 or more days of opioid use in a 28-day period as assessed by self-report or by testing of urine samples obtained every 2 weeks, positive or missing sample imputed as 5 days of opioid use.
Participants Completed | 26 weeks
  Proportion of enrolled participants who complete the intervention period (i.e., do not withdraw consent or are otherwise removed from the study prior to the intervention end date.

CONTACTS AND LOCATIONS:
Locations (1):
- Maryland Treatment Centers, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
After deidentification, the IPD related to primary and secondary outcomes will be made publicly available as required by NIDA data sharing policies.

REFERENCES:
- [Background] Wenzel K, Fishman M. Mobile van delivery of extended-release buprenorphine and extended-release naltrexone for youth with OUD: An adaptation to the COVID-19 emergency. J Subst Abuse Treat. 2021 Jan;120:108149. doi: 10.1016/j.jsat.2020.108149. Epub 2020 Sep 24. PMID 33303086
- [Background] Fishman M, Wenzel K, Vo H, Wildberger J, Burgower R. A pilot randomized controlled trial of assertive treatment including family involvement and home delivery of medication for young adults with opioid use disorder. Addiction. 2021 Mar;116(3):548-557. doi: 10.1111/add.15181. Epub 2020 Aug 4. PMID 32621368
- [Background] Fishman M, Wenzel K, Gauthier P, Borodovsky J, Murray O, Subramaniam G, Levy S, Fredyma E, McLeman B, Marsch LA. Engagement, initiation, and retention in medication treatment for opioid use disorder among young adults: A narrative review of challenges and opportunities. J Subst Use Addict Treat. 2024 Nov;166:209352. doi: 10.1016/j.josat.2024.209352. Epub 2024 Mar 16. PMID 38494051
- [Background] Wenzel K, Selby V, Wildberger J, Lavorato L, Thomas J, Fishman M. Choice of extended release medication for OUD in young adults (buprenorphine or naltrexone): A pilot enhancement of the Youth Opioid Recovery Support (YORS) intervention. J Subst Abuse Treat. 2021 Jun;125:108306. doi: 10.1016/j.jsat.2021.108306. Epub 2021 Jan 26. PMID 34016297
- [Background] Wenzel K, Mallik-Kane K, Anderson K, Fishman M. An Assertive Community Intervention to Engage Youth with Opioid Use Disorder and Their Families. Child Adolesc Psychiatr Clin N Am. 2024 Oct;33(4):709-728. doi: 10.1016/j.chc.2024.02.007. Epub 2024 Apr 6. PMID 39277321